CLINICAL TRIAL: NCT04046198
Title: The Effect of Educational Program Based on Professional Values Model on Professional Values Perception and Job Satisfaction in Pediatric Nurses
Brief Title: Professional Values Perception and Job Satisfaction in Pediatric Nurses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Ayla Kaya, Research Assistant, Akdeniz University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AkdUnv
Record Dates: First submitted 2019-08-02; First posted 2019-08-06 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Nursing
Keywords: Professional Values Model; professional values; job satisfaction; pediatric nursing

STUDY DESIGN:
Intervention Model Description: a non-randomized experimental design with pretest and posttest including intervention and control groups
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- İntervention group (Experimental): Nurses working at Akdeniz University Hospital became the intervention group. The nurses who accepted to participate in the study were divided into groups of 5-15 people. Pre-test was applied to nurses who accepted the research. Nurses were given 4-hour group trainings. A booklet on the subject prepared by the researchers was given. Three interim interviews were conducted in the subsequent 3-month period. Six separate posters were posted in the clinics. Weekly reminder messages were sent via WhatsApp. At the end of the third month, post-test data were collected from the nurses.
  Interventions: Other: Educational program
- Control group (Other): The nurses working in the University of Health Sciences Antalya Training and Research Hospital constituted the control group. Pre-test was applied to nurses who accepted the research. Post test applied 3 months later. A booklet on the subject prepared by the researchers was given after the post test. Group training was conducted to nurses.
  Interventions: Other: Educational program

INTERVENTIONS:
Other: Educational program — The Professional Values Education Program was developed in accordance with the Professional Values Model. For nurses in the intervention group program continued for three months. Group training was given before. Then, three individual interviews were conducted. After the post test was applied to the control group, group training was performed.

SUMMARY:
Objective: This study was conducted to determine the effect of the Professional Values Training Program developed in line with Professional Values Model on the perception of professional values and job satisfaction of pediatric nurses.

Method: The study is non-randomized experimental study that measures with pre-test and post-test which includes intervention and control groups. This study was conducted between December 2018 and May 2019. The sample of the study consisted of 40 intervention and 40 control group pediatric nurses. The intervention group group was involved in 12-week-training program which based on the Professional Values Model. Data were collected by using the Individual Identification Form, the Nurses' Professional Values Scale (NPVS-R) and the Healthcare Environment Survey (HES).

DETAILED DESCRIPTION:
This study was conducted in non-randomized experimental design with pretest and posttest including intervention and control groups to determine the effect of the Professional Values Educational Program developed in accordance with Professional Values Model to test a theoretical model on professional value perception, job satisfaction levels and parental care satisfaction of pediatric nurses.

Pediatric nursing is a field that takes children and families at central point of care and is responsible for providing health care from the neonatal period to the end of adolescence. Pediatric nurses' awareness of professional values is an important issue that should be addressed for development of nursing practices, quality nursing care, professional identity acquisition, high job satisfaction and minimization of leave of employment. In the studies, it is reported that the development of professional values is an important factor that increases the satisfaction of individuals receiving care and the job satisfaction of nurses.

Ethics committee approval and written permission were obtained from the hospitals before the study was conducted. Written consent was obtained from all participating nursesIn the study. Personal Information Form, Nursing Professional Values Scale (NPVS-R) and Healthcare Environment Survey (HES) were used as data collection tools. These data collection tools were used in the pre-test and post-test.

Nurses working at Akdeniz University Hospital became the intervention group. The nurses who accepted to participate in the study were divided into groups of 5-15 people. Pre-test was applied to nurses who accepted the research. Nurses were given four group trainings. A booklet on the subject prepared by the researchers was given. Three interim interviews were conducted in the subsequent 12-week. Six separate posters were posted in the clinics. Weekly reminder messages were sent via WhatsApp. At the end of the third month, post-test data were collected from the nurses.

The nurses working in the University of Health Sciences Antalya Training and Research Hospital constituted the control group. Pre-test was applied to nurses who accepted the research. Post test applied 3 months later. A booklet on the subject prepared by the researchers was given after the post test. Group training was conducted to nurses.

The post test data was collected in May 2019.

ELIGIBILITY:
Inclusion Criteria:

- Being a nurse directly responsible for the care of the child patient

Exclusion Criteria:

* Failure to complete the Professional Values Training Program
* Want to leave the research
* Leave the clinic for any reason / relocation / dismissal, etc.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-12-21 (Actual); Primary Completion 2019-01-17 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
Nurses' Professional Values Scale (NPVS-R) | Three months
  The Nurses' Professional Values Scale was developed by Weis & Schank in 2000. Validity and reliability Geçkil et al. (2012) did in Turkey. The scale has a total of 26 items. Each item is scored from 1 to 5. The lowest score that can be obtained from the total scale is 26 and the highest score is 130. The higher the total score, the more important the professional values of nurses. The pre-test and post-test data of the intervention group and control group will be analyzed. The 3-months education program was applied only to the intervention group. Therefore, there is no success criteria in the control group. The statistically significant increase in the mean score of professional values in posttest measurement in the intervention group is the success criterion of the study. Significance level is set at p<0.05 in analyzes.
Healthcare Environment Survey (HES) | Three months
  The Health Environment Survey was developed in 2001 to assess the job satisfaction of nurses. It was revised in 2015 (Nelson et al., 2015). Gözüm, Nelson, Yıldırım & Kavla, (2017) adapted the scale into the Turkish culture and found the scale as valid and reliable. The scale has a total of 61 items. Each item is scored from 1 to 7. By adding the points and dividing them by the number of items, the scale score averages are obtained. Neutral point average of 3.5. The higher the average score, the higher the job satisfaction. The survey measures 11 dimensions of nurse job satisfaction. At the end of the 3-months education program, it was expected that job satisfaction scores would increase significantly in the intervention group. The statistically significant increase in the mean score of job satisfaction in posttest measurement in the intervention group is the success criterion of the study. Significance level is set at p<0.05 in analyzes.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşegül İŞLER DALGIÇ, Professor, Study Director — Akdeniz University
Locations (1):
- Ayla Kaya, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kaya A, Boz I. The development of the Professional Values Model in Nursing. Nurs Ethics. 2019 May;26(3):914-923. doi: 10.1177/0969733017730685. Epub 2017 Sep 20. PMID 28929939
- [Background] Kantek F, Kaya A. Professional Values, Job Satisfaction, and Intent to Leave Among Nursing Managers. J Nurs Res. 2017 Aug;25(4):319-325. doi: 10.1097/JNR.0000000000000164. PMID 28683021
- [Background] Geckil E, Ege E, Akin B, Goz F. Turkish version of the revised nursing professional values scale: validity and reliability assessment. Jpn J Nurs Sci. 2012 Dec;9(2):195-200. doi: 10.1111/j.1742-7924.2011.00202.x. Epub 2012 Jan 18. PMID 23181888
- [Background] Yarbrough S, Martin P, Alfred D, McNeill C. Professional values, job satisfaction, career development, and intent to stay. Nurs Ethics. 2017 Sep;24(6):675-685. doi: 10.1177/0969733015623098. Epub 2016 Jan 24. PMID 26811397
- [Background] Weis D, Schank MJ. Development and Psychometric Evaluation of the Nurses Professional Values Scale-3. J Nurs Meas. 2017 Dec 1;25(3):400-410. doi: 10.1891/1061-3749.25.3.400. PMID 29268825
- [Background] Roney LN, Acri MC. The Cost of Caring: An Exploration of Compassion Fatigue, Compassion Satisfaction, and Job Satisfaction in Pediatric Nurses. J Pediatr Nurs. 2018 May-Jun;40:74-80. doi: 10.1016/j.pedn.2018.01.016. Epub 2018 Feb 3. PMID 29402658
- [Background] Akman O, Ozturk C, Bektas M, Ayar D, Armstrong MA. Job satisfaction and burnout among paediatric nurses. J Nurs Manag. 2016 Oct;24(7):923-933. doi: 10.1111/jonm.12399. Epub 2016 Jun 7. PMID 27271021